CLINICAL TRIAL: NCT03956771
Title: Neurofeedback With Magnetic Resonance Imaging (MRI) for OCD Participants With Treatment-resistance
Brief Title: Neurofeedback for Treatment-resistant Obsessive-compulsive Disorder (OCD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pedro Morgado (Other)
Collaborators: Hospital de Braga (Other); Clinical Academic Center (2CA) (Unknown)
Responsible Party: Sponsor-Investigator, Pedro Morgado, Assistant Professor, M.D., Ph.D., University of Minho
Organization: University of Minho (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OCDNF_ICVS2019
Record Dates: First submitted 2019-05-16; First posted 2019-05-21 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Obsessive-Compulsive Disorder; OCD
Keywords: neurofeedback; biofeedback; OCD; obsessive-compulsive disorder; magnetic resonance imaging; functional magnetic resonance imaging; orbitofrontal cortex
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Intervention Model Description: OCD participants will be blindly split into two groups (n = 15): the real neurofeedback group (group 1, experimental group) and the sham neurofeedback group (group 2, sham comparator control group). Group 1 will receive feedback information from real activity from the target brain region, while group 2 will receive false feedback not matching real brain responses to account for placebo effects (from other participant's data).
Who Masked: Participant, Outcomes Assessor
Masking Description: OCD participants will be blindly split into the two groups before the neurofeedback intervention. The psychologist evaluating the psychometric outcomes will be blind to the type of intervention of each participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real neurofeedback (Experimental): Two sessions of neurofeedback training during 2 weeks (2 distinct days; 36 min per session).
  Interventions: Behavioral: Real neurofeedback
- Sham neurofeedback (Sham Comparator): Two sessions of placebo/control neurofeedback training during 2 weeks (2 distinct days; 36 min per session).
  Interventions: Behavioral: Sham neurofeedback

INTERVENTIONS:
Behavioral: Real neurofeedback — Regulation of brain activity in real-time with feedback from brain activity measured with MRI from the orbitofrontal cortex of the participant him/herself. Participants receive feedback of their own brain activity in a screen with pictures. Participants are instructed to try to decrease the pictures transparency to reduce the orbitofrontal cortical activity. Psychotherapy strategies to decrease brain responses will be teach to the participants before the intervention.
  Arms: Real neurofeedback
Behavioral: Sham neurofeedback — Regulation of brain activity in real-time with feedback from brain activity measured with MRI from the orbitofrontal cortex of other participant. Participants receive feedback of other participant' brain activity in a screen with pictures. Participants are instructed to try to decrease the pictures transparency to reduce the orbitofrontal cortex activity. Psychotherapy strategies to decrease brain responses will be teach to the participants before the intervention.
  Arms: Sham neurofeedback

SUMMARY:
The aim of this study is to teach participants with a OCD diagnosis and treatment-resistance how to decrease the response from a brain region involved in the disease by using a technique called neurofeedback. While using this technique, the participants visualize their own brain response in a screen during a MRI exam. Participants will learn strategies to decrease brain responses. The neurofeedback technique is non-invasive, without known risks to participants. With this study, it is expect that the neurofeedback training over 2 weeks (2 sessions) will reduce the OCD symptoms when compared to a control intervention based on neurofeedback's placebo effects.

DETAILED DESCRIPTION:
OCD individuals will be recruited at Hospital of Braga, Braga, Portugal, in collaboration with the Psychiatry Unit (n = 30, nonrandom convenience sample based on effect size of 0.30, alpha = beta = 0.05, and ANOVA repeated measures within-between interaction). Some participants may quit the study but sample size was predetermined considering a putative 30 percent dropout rate. Clinical history will be assessed (sociodemographic information, disease onset and severity, and previous/current treatments). The participants' neuropsychological state, the blood hormonal levels, and brain function and structure as baseline measures before and after the neurofeedback intervention will be assessed. Two MRI neurofeedback sessions will be performed during 2 weeks (2 distinct days; 36 min per session) in a 3 T MRI scanner. Data analysis will be performed with a repeated measures design (baseline and after neurofeedback) between the groups to measure brain, blood, and neuropsychological changes. Patients will be supervised by a physician to track putative complications/adverse effects during the intervention. The participation will be immediately interrupted in case of adverse reactions or symptomatic worsening and a physician will follow the participants to provide the appropriated care.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of current OCD according to the fifth Diagnostic and Statistical Manual of Mental Disorders;
* Treatment resistance (≥ 3 selective serotonin reuptake inhibitors in proper dose for ≥ 12 weeks).

Exclusion Criteria:

* Concomitant psychiatric or neurological illness;
* Substance abuse/dependence in the past 6 months (except nicotine/caffeine);
* Acute suicidal ideation;
* Psychotropic medication (except selective serotonin reuptake inhibitors, anafranil, or low-dose hypnotic or anxiolytic taken occasionally);
* MRI contraindications (pregnancy, major head trauma, severe claustrophobia, severe back pain, ferromagnetic materials/prostheses/implants inside the body, or other).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-04-05 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline in Yale-Brown Obsessive Compulsive Scale score. | 2-3 days before the intervention, 2-3 days after the intervention, and 3 months after the intervention.
  Psychometric scale to evaluate obsessive-compulsive symptoms. The total score ranges from 0 to 50 with the following classification: 0-7 sub-clinical symptoms, 8-15 moderate symptoms, 16-31 severe symptoms, and >= 32 extreme symptoms. This scale can be divided into two subscales: compulsions subscale (score ranging from 0 to 25) and obsessions subscale (score ranging from 0 to 25). The sum of the subscales scores gives the total score of the scale. Lower total and subscale scores represent a better outcome.
Mean change from baseline in Obsessive-Compulsive Inventory-Revised score. | 2-3 days before the intervention, 2-3 days after the intervention, and 3 months after the intervention.
  Psychometric scale to evaluate obsessive-compulsive symptoms. The total score ranges from 0 to 72. This scale can be divided into six subscales: checking subscale (score ranging from 0 to 12), hoarding subscale (score ranging from 0 to 12), neutralizing subscale (score ranging from 0 to 12), obsessing subscale (score ranging from 0 to 12), ordering subscale (score ranging from 0 to 12), and washing subscale (score ranging from 0 to 12). The sum of the subscales scores gives the total score of the scale. Lower total and subscale scores represent a better outcome.
Mean change from baseline in Hamilton Anxiety Rating Scale score. | 2-3 days before the intervention, 2-3 days after the intervention, and 3 months after the intervention.
  Psychometric scale to evaluate anxiety symptoms. The total score ranges from 0 to 56 with the following classification: 0-16 mild anxiety symptoms, 17-24 mild to moderate anxiety symptoms, 25-30 moderate to severe anxiety symptoms, and >= 31 severe anxiety symptoms. Lower total scores represent a better outcome.
Mean change from baseline in Hamilton Depression Rating Scale score. | 2-3 days before the intervention, 2-3 days after the intervention, and 3 months after the intervention.
  Psychometric scale to evaluate depression symptoms. The total score ranges from 0 to 52 with the following classification: 0-7 no symptoms, 8-16 mild depression symptoms, 17-23 moderate depression symptoms, and >= 24 severe depression symptoms. Lower total scores represent a better outcome.
Mean change from baseline in State-Trait Anxiety Inventory score. | 2-3 days before the intervention, 2-3 days after the intervention, and 3 months after the intervention.
  Psychometric scale to evaluate anxiety symptoms. The total score ranges from 40 to 160 with the following classification: 40-76 sub-clinical symptoms, >= 78 clinical symptoms. This scale can be divided into two subscales: state anxiety subscale (score ranging from 20 to 80) and trait anxiety subscale (score ranging from 20 to 80). The sum of the subscales scores gives the total score of the scale. Lower total and subscale scores represent a better outcome.
Mean change from baseline in the score of Perceived Stress Scale with 10 items. | 2-3 days before the intervention, 2-3 days after the intervention, and 3 months after the intervention.
  Psychometric scale to evaluate perceived stress symptoms. The total score ranges from 0 to 40. Lower total scores represent a better outcome.
Mean change from baseline in Emotion Regulation Questionnaire score. | 2-3 days before the intervention, 2-3 days after the intervention, and 3 months after the intervention.
  Psychometric scale to evaluate cognitive regulation and emotional suppression capabilities. The cognitive regulation subscale score ranges from 6 to 42 and the emotional suppression subscale score ranges from 4 to 28. Lower emotional suppression scores and higher cognitive regulation scores represent a better outcome.

SECONDARY OUTCOMES:
Difference from baseline in functional connectivity patterns in the brain. | 2-3 days before the intervention, 2-3 days after the intervention
  Functional connectivity maps will be obtained with resting state functional MRI sequences to study changes in brain function induced by the intervention, mainly in regions associated with the target region - the orbitofrontal cortex.
Differences from baseline in brain grey and white matter structure. | 2-3 days before the intervention, 2-3 days after the intervention
  Diffusion tensor imaging and anatomical MRI sequences will be applied to assess brain white matter integrity and gray matter morphology, respectively.
Mean change from baseline in blood hormonal composition | 2-3 days before the intervention, 2-3 days after the intervention
  Hemogram and measurement of thyroid-stimulating hormone, cortisol, glucose, and adrenocorticotropic hormone levels in the blood.

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Morgado, M.D., Ph.D., Principal Investigator — Life and Health Sciences Research Institute (ICVS), School of Medicine, University of Minho; ICVS/3B's - PT Government Associate Laboratory; Braga, Portugal
Locations (1):
- Life and Health Sciences Research Institute, School of Medicine, University of Minho, Braga, Gualtar, Portugal

IPD SHARING:
Plan to Share IPD: No